CLINICAL TRIAL: NCT00686088
Title: An Open-Label, Multi-Center, Phase IIa Trial of PRX302 Treatment of Patients With Locally Recurrent Prostate Cancer After Primary Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sophiris Bio Corp (Industry)
Responsible Party: Rosemina Merchant, M.E.Sc., VP, Development and Regulatory Affairs, Protox Therapeutics
Organization: Protox Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRX302-1-02
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-09

CONDITIONS: Locally Recurrent Prostate Cancer
Keywords: prostate cancer; locally recurrent; PRX302
MeSH Terms: conditions — Prostatic Neoplasms | interventions — PRX302

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PRX302 — Determination of the therapeutic activity of different concentrations of PRX302 at increasing volumes and/or number of deposits per gram of prostate.

SUMMARY:
The purpose of this study is to determine the therapeutic activity of different concentrations of PRX302 at increasing volumes and/or number of deposits per gram of prostate. Therapeutic activity will be determined based on changes in PSA levels, PSA velocity, PSA doubling time and tumor burden following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Completed a full course of radiation therapy for prostate cancer at least 2 years before enrollment.
* Biochemical failure at screening as determined by either the ASTRO or the Phoenix definitions.
* At least 5 available PSA readings after completion of radiation therapy and prior to screening.
* PSA level of not greater than 10 ng/mL.
* PSA doubling time of at least 9 months at screening.
* Biopsy-proven recurrent localized prostate cancer.
* Tumor stage T1C to T2C.
* Prostate volume estimated at 40 mL or less as determined by TRUS.
* ECOG performance score 0 to 2.
* Serum testosterone of at least 1 ng/dL.

Exclusion Criteria:

* Prior history of metastatic prostate cancer.
* Salvage external beam therapy and/or salvage brachytherapy prior to enrollment.
* Biological, immunological, chemotherapeutic treatment or cryotherapy after completing radiation.
* Androgen ablation therapy within 12 months prior to enrollment.
* Recurrence of prostate cancer within 18 months of definitive primary radiotherapy.
* Other medication for prostate cancer.
* Presence of active malignancy other than prostate cancer.
* Treatment with other investigational therapies within 12 months prior to enrolment.
* Presence of a chronic indwelling Foley catheter for obstructive uropathy.
* Previous transurethral resection of the prostate (TURP), transurethral resection of the bladder neck, photo-selective vaporization of the prostate (PVP) or other resection surgery in the urinary tract.
* Previous treatment with PRX302.
* Any evidence of metastatic disease on bone scan, CT or magnetic resonance imaging (MRI) within 3 months prior to enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
PSA levels, PSA doubling time, PSA velocity and tumor burden assessment by biopsy compared to screening. | Day 45 and Day 180

SECONDARY OUTCOMES:
Safety and tolerability of PRX302. | 12 months.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Urology San Antonio, San Antonio, Texas
  - Scott & White Memorial Hospital, Temple, Texas